CLINICAL TRIAL: NCT06393985
Title: A Multicenter, Prospective, Phase II Study of Decitabine, Venetoclax and Blinatumomab for Maintenance Following Allogeneic Hematopoietic Cell Transplantation in Patients With Ph-Negative B-Cell Acute Lymphoblastic Leukemia
Brief Title: Decitabine, Venetoclax and Blinatumomab for Maintenance Following HSCT in Patients With Ph-Negative B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstSoochowU-DVB
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-04

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Ph-negative B-ALL; HSCT; maintenance therapy
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Decitabine; venetoclax; blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decitabine,venetoclax and blinatumomab (Experimental)
  Interventions: Drug: Decitabine, venetoclax and blinatumomab

INTERVENTIONS:
Drug: Decitabine, venetoclax and blinatumomab — Cycle1 and cycle3： Decitabine monotherapy,20 mg/m2 qd, d1-5,intravenous infusion;
  Cycle2 and cycle4:
  Venetoclax 200mg qd, d1-14, orally; Blinatumomab d4-17(Weight ≥45 kg, 9ug d4-6, 28ug d7-17; Weight <45 kg, 5ug/m2 d4-6, 15ug/m2 d7-17;continuous intravenous infusion)

SUMMARY:
This study aims to evaluate whether maintenance therapy with decitabine, venetoclax and blinatumomab could improve the 2-year progression free survival (PFS) of patients with philadelphia chromosome-negative B-cell acute lymphoblastic leukemia who had recently received an allogeneic stem cell transplant and in measurable residual disease-negative remission.

DETAILED DESCRIPTION:
This is a phase Ⅱ, open-label, single-arm, multi-center study in patients with philadelphia chromosome-negative B-cell acute lymphoblastic leukemia who had recently received an allogeneic stem cell transplant and in minimal residual disease-negative remission. In this study, patients will be treated with 4 cycles of maintence therapies for up to one year (or until intolerable toxicity, death, withdrawal, or study termination). In cycle one and three, patients will receive decitabine monotherapy, and in cycle two and four, patients will receive a combination of venetoclax and blinatumomab. This study aims to evaluate whether maintenance therapy with decitabine, venetoclax and blinatumomab could improve the 2-year progression free survival (PFS) of those patients, and explore the efficiency and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1.Philadelphia chromosome-negative B-cell acute lymphoblastic leukemia who underwent an alloHSCT as follows:

  1. patients in CR1 with high-risk features,including adverse clinical features, cytogenetic or molecular alterations according to NCCN 2023.V3.
  2. patients lack of achievement of complete remission after standard induction chemotherapy.
  3. patients with detectable minimal residual disease pre-transplantation.
  4. patients in second and higher CR pre-transplantation. 2.Negative minimal residual disease prior to enrollment (FCM-MRD <0.01% and fusion gene negative).

  3.≥3 months post-transplantation. 4.hematopoietic reconstitution, i.e., ANC ≥0.5 x 109/L, and platelets >20 x 109/L.

  5.Eastern Cooperative Oncology Group (ECOG) score: 0-2. 6.Total serum bilirubin ≤ 3 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 5 x ULN, aspartate aminotransferase (AST) ≤ 5 x ULN.

  7.Creatinine clearance ≥ 30 mL/min. 8.Provide informed consent.

Exclusion Criteria:

* 1.Patients with another malignant disease. 2.Patients with uncontrolled active infection. 3.Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.

  4.Detectable minimal residual disease post-transplantation 5.Active GVHD requiring systemic steroid therapy. 6.Patients with uncontrolled active bleeding. 7.Pregnant and lactating women; patients of childbearing potential should be willing to practice methods of contraception throughout the study period.

  8.Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of allogenetic HSCT until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after allogenetic HSCT
  Progression-free survival (PFS) was defined as the period from the date of allogenetic HSCT to the observed progression of the disease or the occurrence of death for any reason.(Progression is defined as more than 5% blast in the peripheral blood or bone marrow biopsy.)

SECONDARY OUTCOMES:
OS | 2 years after allogenetic HSCT
  Overall survival (OS) is defined as the period from the date of allogenetic HSCT to the date of death.
CIR | 2 years after allogenetic HSCT
  Cumulative incidence of relapse（CIR）is measured from the date of achievement of remission until the date of hematologic relapse, or MRD relapse. Patients who died without relapsing are counted as a competing cause of failure.
TEAE | From the start of each cycle to 30 days after the end
  Treatment-emergent adverse event (TEAE; frequency, CTCAE grade） is defined as an AE observed after starting administration of the study treatment until 30 days from the end.
GRFS | 2 years after allogenetic HSCT
  GVHD-free relapse-free survival (GRFS) is defined as the time from the date of allogenetic HSCT until the date of treatment-emergent acute GVHD III-IV, or treatment-emergent chronic GVHD that requires new or additional immunosuppressive treatment, or morphological relapse or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No